CLINICAL TRIAL: NCT03428243
Title: Long-term Follow-up Study of the truSculpt Radiofrequency Device for Circumferential Reduction: 18-month Circumference Measuing of Some C-16-TS11 Subjects.
Brief Title: Long-term Follow-up Study of the truSculpt Radiofrequency Device for Circumferential Reduction
Status: Completed | Type: Observational
Sponsor: Cutera Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: C-17-TS15
Record Dates: First submitted 2018-02-05; First posted 2018-02-09 (Actual); Last update posted 2018-03-20 (Actual); Status verified 2018-02

CONDITIONS: Abdominal Fat

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- truSculpt: truSculpt effectiveness after 18 months
  Interventions: Device: truSculpt

INTERVENTIONS:
Device: truSculpt — Device comparison of Circumference measurement at Baseline vs 18 months post treatment

SUMMARY:
A long-term follow-up study to evaluate the safety and efficacy of the Cutera truSculpt radiofrequency device for circumferential reduction.

DETAILED DESCRIPTION:
The purpose of this investigation is to follow-up subjects who have completed participation in the Treatment Group of Protocol C-16-TS11 - "Pivotal Study of the TruSculpt Radiofrequency Device for Circumferential Reduction" for the long-term (18 months) safety and efficacy of the truSculpt radiofrequency (RF) device for circumferential reduction in the abdominal and flank region.

ELIGIBILITY:
Inclusion Criteria:

1. Completed participation in the Treatment Group of Protocol C-16-TS11 - "Pivotal Study of the TruSculpt Radiofrequency Device for Circumferential Reduction"
2. Subject has maintained the same weight since enrolling in Protocol C-16-TS11 - "Pivotal Study of the TruSculpt Radiofrequency Device for Circumferential Reduction", within 5% of baseline weight measurement.

Exclusion Criteria:

1. Participation in a clinical trial of another device or drug in the target area since enrolling in Protocol C-16-TS11 - "Pivotal Study of the TruSculpt Radiofrequency Device for Circumferential Reduction".
2. Any type of cosmetic treatment to the target area to reduce circumference since enrolling in Protocol C-16-TS11 - "Pivotal Study of the TruSculpt Radiofrequency Device for Circumferential Reduction" e.g., radiofrequency, cryolysis or light-based treatments.
3. Any invasive cosmetic surgery to the target area, such as liposuction, since enrolling in Protocol C-16-TS11 - "Pivotal Study of the TruSculpt Radiofrequency Device for Circumferential Reduction".
4. Newly diagnosed (since enrolling in Protocol C-16-TS11) significant concurrent illness, such as diabetes mellitus, cardiovascular disease, peripheral vascular disease or pertinent neurological disorders.
5. Newly diagnosed or documented (since enrolling in Protocol C-16-TS11) immune system disorders.
6. Current infection, dermatitis, rash or other skin abnormality in the treatment area.
7. Currently undergoing systemic chemotherapy or radiation treatment for cancer, or treatment in the target area since enrolling in Protocol C-16-TS11 - "Pivotal Study of the TruSculpt Radiofrequency Device for Circumferential Reduction".
8. Pregnant or currently breastfeeding.
9. As per the Investigator's discretion, any physical or mental condition which might make unsafe for the subject to participate in this study.

Ages: 24 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 14 Subjects from C-16-TS11 participants followed up for measurement
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2017-07-12 (Actual); Primary Completion 2017-11-06 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
Circumference Measurement | 18 months post C-16-TS11 completion (September, 2016)
  Comparison of Abdominal region Measurement in cm 18 months post-treatment with C-16 TS11 Baseline.

SECONDARY OUTCOMES:
Device Safety | 18 months post C-16-TS11 completion (September, 2016)
  Measurement of Resolved Adverse Events from Radiofrequency (RF) treatment (C-16-TS11), and Presence of any Additional AE within 18 months of RF treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Ronan, MD, Principal Investigator — Principal Investigator
Locations (1):
- Cutera Research Center, Brisbane, California, United States